CLINICAL TRIAL: NCT05708599
Title: Longitudinal Liquid Biopsy Study Without an Investigational Medicinal Product in Patients With Non-Small Cell Lung Cancer (NSCLC) Including Squamous Cell Carcinoma, Adenocarcinoma and Large Cell Carcinoma, Colorectal Carcinoma (CRC) and Pancreatic Ductal Adenocarcinoma (PDAC) to Evaluate Novel Blood-based Biomarkers for Use in Early Clinical Development
Brief Title: A Study to Compare Tissue and Liquid Biopsies in People With Different Types of Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Universitätsklinikum Kiel, Onkologisches Zentrum (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0352-2187
Record Dates: First submitted 2023-01-16; First posted 2023-02-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-Small-Cell Lung Carcinoma; Colorectal Cancer; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with early-stage and advanced-stage disease per indication (Experimental): Indications: Pancreatic ductal adenocarcinoma (PDAC), colorectal carcinoma (CRC) and non-small cell lung cancer (NSCLC)
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — Liquid biopsy

SUMMARY:
In study, liquid biopsy samples will be obtained from non-small cell lung cancer (NSCLC) including Squamous cell carcinoma, Adenocarcinoma and large cell carcinoma, colorectal carcinoma (CRC) and pancreatic ductal adenocarcinoma (PDAC) patients who undergo treatment according to established standards of care (SoC) at the University Hospital Schleswig-Holstein (UKSH).

This study will observe the overall Variant Allele Frequency (VAF) of circulating tumour Desoxyribonucleic acid (ctDNA) levels over the patient therapeutic treatment course and will correlate these findings with tumour response as well as Kirsten rat sarcoma viral oncogene homolog (KRAS)mutation status.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Male or female patients with pancreatic ductal adenocarcinoma, colorectal carcinoma or adenocarcinoma of the lung as specified above leading to new treatment line.
3. Signed and dated written informed consent in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the study.
4. Willingness to undergo pre- and on-treatment liquid biopsies for biomarker assessment. Patients can be enrolled without tissue tumour biopsy upon agreement between the Investigator and the Sponsor.

Exclusion Criteria:

1. Patients not expected to comply with the protocol requirements or not expected to complete the study as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable study participant).
2. Women who are pregnant or who plan to become pregnant during the study.
3. Participation at a clinical trial involving an investigational medicine where the treatment details cannot be disclosed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-02-08 (Estimated); Study Completion 2027-02-08 (Estimated)

PRIMARY OUTCOMES:
Mean variant allele frequency (VAF) of mutations in circulating tumour Desoxyribonucleic acid (ctDNA) samples over the timescale of the patient's treatment course | up to 5 years

SECONDARY OUTCOMES:
Tumour growth/tumour marker changes for each therapeutic treatment regimen at each biopsy sampling time point as compared to baseline | up to 5 years
Correlation of Kirsten rat sarcoma viral oncogene homolog (KRAS) mutation status and objective response | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com